CLINICAL TRIAL: NCT00612859
Title: A Multicenter, Randomized, Double-Blind, PBO-Controlled, Parallel Group Study to Assess the Efficacy and Safety of Levetiracetam Versus PBO for the Treatment of Social Anxiety Disorder (Generalized Type)
Brief Title: Study to Assess the Efficacy and Safety of Levetiracetam for the Treatment of Social Anxiety Disorder (Generalized Type)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01086
Record Dates: First submitted 2008-01-14; First posted 2008-02-12 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2009-09

CONDITIONS: Anxiety Disorders
Keywords: Levetiracetam; Keppra
MeSH Terms: conditions — Anxiety Disorders | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: levetiracetam

SUMMARY:
Preclinical and clinical findings indicate that LEV has some anxiolytic potential. There is reason to believe that compounds with anxiolytic activity may have broad clinical utility across the anxiety spectrum. This trial was intended to explore LEV's utility in adults with social anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients between 18 and 70 years old inclusive;
* symptoms of social anxiety disorders (generalized type) present for at least 1 year prior to Selection Visit;
* had a score of >=60 on the LSAS at the Selection Visit and at the Randomization Visit. Additionally, the clinician's gloal impression of change score must have been >= 2 at the Randomization Visit;
* had a telephone where they could be directly contacted.

Exclusion Criteria:

* History of autism or Asperger's Disease;
* had another primary axis I disorder or fulfilled diagnostic and statistical manual of mental disorders-4th edition (DSM-IV) criteria in the 6 months prior to Screening;
* major depression as measured by a Hamilton Depression Rating Scale (HAM-D-17 items) total score of > 17 and/or a suicide subscale score on the HAM-D-17 items of > 2 at the Selection or Randomization Visit;
* history of electroconvulsive therapy within the prior 3 months;
* history of psychotherapy which was not stable and ongoing for at least 6 months prior to Visit 1;
* clinical history of significantly impaired renal function with an estimated creatinine clearance below 80 mL/min;
* clinically significant medical condition;
* history of any clinically significant allergic condition or allergy to LEV or pyrrolidone derivatives;
* neutrophil count of less than 1800/µL.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2003-09; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
change in Liebowitz Social Anxiety Scale (LSAS) score from Visit 2 to the last Evaluation period visit attended using last observation carried forward (LOCF) methods
Safety: monitoring of AEs, clinical laboratory tests, physical examination and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)